CLINICAL TRIAL: NCT02507765
Title: A Pilot Trial of Stereotactic Body Radiation Therapy (SBRT) to Induce Tumor Hyperemia in Combination With Transarterial Chemoembolization (TACE) for Unresectable Hepatocellular Carcinoma
Brief Title: Stereotactic Body Radiation Therapy and Transarterial Chemoembolization in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-15032; NCI-2015-00894 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Child-Pugh Class A; Child-Pugh Class B; Stage IIIA Hepatocellular Carcinoma; Stage IIIB Hepatocellular Carcinoma; Stage IIIC Hepatocellular Carcinoma; Stage IVA Hepatocellular Carcinoma; Stage IVB Hepatocellular Carcinoma
Keywords: SBRT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SBRT, TACE) (Experimental): Patients undergo SBRT on day 1 and TACE on day 2.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Stereotactic Body Radiation Therapy; Procedure: Transarterial Chemoembolization

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SBRT
Procedure: Transarterial Chemoembolization — Undergo TACE
  Other Names: TACE

SUMMARY:
This pilot clinical trial studies stereotactic body radiation therapy (SBRT) and transarterial chemoembolization (TACE) in treating patients with liver cancer that cannot be removed by surgery. SBRT is a specialized radiation therapy that delivers a high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue. Chemoembolization kills tumor cells by carrying drugs directly into blood vessels near the tumors and then blocking the blood flow to allow a higher concentration of the drug to reach the tumor for a longer period of time. SBRT may make TACE more beneficial by increasing blood flow to the tumor, which may allow more of the TACE chemotherapy to enter the tumor. Giving SBRT with TACE may work better in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the feasibility of completing SBRT followed by TACE in a 2 day time period.

SECONDARY OBJECTIVES:

I. To determine acute tumor perfusion changes after SBRT using functional magnetic resonance imaging (MRI) (magnetic resonance [MR]-dynamic contrast enhanced [DCE]/perfusion weighted imaging [PWI], MR-diffusion, blood oxygen level dependent [BOLD] sequences).

II. To establish safety and tolerability of this regimen. III. To determine overall response rates (using modified Response Evaluation Criteria in Solid Tumors [RECIST] criteria), including objective response rate (partial response [PR] + complete response [CR]) and clinical benefit rate (stable disease [SD] + PR + CR) at 1, 3, and 6 months after TACE.

IV. To evaluate local control, progression-free survival, and overall survival at 1, 3, 6, 9, and 12 months after a single-dose of SBRT followed by TACE.

V. To correlate micro ribonucleic acid (miRNA) biomarkers with response and toxicity.

OUTLINE: This is a dose-escalation study of SBRT.

Patients undergo SBRT on day 1 and TACE on day 2.

After completion of study treatment, patients are followed up at 1-2 weeks and at 1, 3, 6, 9, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of hepatocellular carcinoma by at least one criterion listed below:

  * Histologically confirmed
  * Magnetic resonance imaging (MRI) or computerized tomography (CT) findings consistent with hepatocellular carcinoma
  * Alpha fetoprotein (AFP) > 400 ng/mL AND evidence of at least one solid liver lesion > 2 cm regardless of specific imaging characteristics on CT or MRI
* Patients must be non-transplantable, unresectable, or medically inoperable and eligible for TACE as determined by a multi-disciplinary team
* Absolute neutrophil count >= 1.5 × 10^9/L
* Hemoglobin >= 9 g/dl
* Platelets >= 50,000/mm^3
* Prothrombin time (PT)/international normalized ratio (INR) and activated partial thromboplastin time (PTTa) =< 1.5
* Albumin >= 2.5 g/dL
* Alkaline phosphatase < 5 x upper limit of normal (ULN)
* Total bilirubin =< 2.0 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x ULN
* Creatinine =< 1.5 mg/dL and calculated creatinine clearance >= 60 mL/min or 24-hour urine creatinine clearance >= 60 mL/min
* Must have Childs-Pugh A or B liver disease
* Patients must have no clinical signs of heart failure and meet New York Heart Association functional classification I or II defined as:

  * Class I - patients with no limitation of activities; they suffer no symptoms from ordinary activities
  * Class II - patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion
* Must have 1-3 liver lesions amenable to SBRT with tumor size < 15 cm (single lesion or sum)
* Must be able to undergo two MRI scans, one before study treatment begins and another shortly after SBRT
* Patients with extrahepatic disease, portal hypertension, or bilobar disease are allowed
* Normal renal function (creatinine < 1.5 mg/dL)
* Within 2 weeks of registration: patients must have vital signs, history/physical examination, laboratory studies (complete blood count [CBC] with differential, chemistries including liver function tests, AFP, creatinine clearance [CrCl] assessment, pregnancy test if needed)
* Life expectancy of at least 12 weeks in the opinion of investigator
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test within 14 days of the first administration of study treatment; urine human chorionic gonadotropin (HCG) is an acceptable pregnancy assessment
* Women/men of reproductive potential must be counseled on contraception/abstinence while receiving the study treatment

Exclusion Criteria:

* Childs-Pugh C liver function
* Major liver vascular invasion
* Prior radiation to the liver or other upper abdominal regions
* Must not have any evidence of bleeding diathesis or active gastrointestinal bleeding
* Any concurrent malignancy other than non-melanoma skin cancer, non-invasive bladder cancer, or carcinoma in situ of the cervix; patients with a previous malignancy without evidence of disease for >= 3 years will be allowed to enter the trial
* History of active connective tissue disease (scleroderma)
* Subjects who are breast-feeding, or have a positive pregnancy test will be excluded from the study; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Medical contraindication to MR imaging (e.g. pacemakers, metallic implants, aneurysm clips, known contrast allergy to gadolinium contrast, pregnancy, nursing mothers, weight greater than 350 pounds)
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the investigator; this could include severe, active co-morbidities such as:

  * Uncontrolled cardiac disease (hypertension, unstable angina, myocardial infarction within last 6 months, uncontrolled congestive heart failure, cardiomyopathy with decreased ejection fraction)
  * Acute bacterial or fungal infection requiring intravenous antibiotics at time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
  * Hepatic insufficiency resulting in jaundice and/or coagulation defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of SBRT in combination with TACE, measured by the number of patients able to tolerate all study procedures | 2 days
  Determined on the intent-to-treat principle. Any treatment delivery difficulties that arise that could impede successful delivery of this therapy sequence will be evaluated. The capability of the Ohio State University (OSU) system and communication between departments will be analyzed and deemed effective if it facilitates the successful treatment completion of all patients.

SECONDARY OUTCOMES:
Change in diffusion | Baseline to day 1 post-SBRT
  Tested by comparing mean values pre- and post-SBRT using a paired t-test. Should there be concern for outliers, the median for each metric will be determined and compared using a corresponding non-parametric procedure.
Change in hypoxia measurements | Baseline to day 1 post-SBRT
  Tested by comparing mean values pre- and post-SBRT using a paired t-test. Should there be concern for outliers, the median for each metric will be determined and compared using a corresponding non-parametric procedure.
Change in perfusion | Baseline to day 1 post-SBRT
  Tested by comparing mean values pre- and post-SBRT using a paired t-test. Should there be concern for outliers, the median for each metric will be determined and compared using a corresponding non-parametric procedure.
Incidence of toxicities | Up to 30 days
  Includes measurement of grade 2-5 gastrointestinal symptoms, such as nausea, abdominal pain, hepatitis, enteritis, gastritis, bowel perforation, and fistula, as defined by Common Terminology Criteria for Adverse Events version 4.03.
Local control | Up to 12 months
  Calculated using standard clinical follow-up with MRI imaging and labs.
Objective response rate (CR + PR) as measured by modified RECIST criteria version 1 | Up to 6 months
Overall survival | Up to 12 months
  Calculated using standard clinical follow-up with MRI imaging and labs. Estimated using Kaplan-Meier analysis.
Progression-free survival | Up to 12 months
  Calculated using standard clinical follow-up with MRI imaging and labs. Estimated using Kaplan-Meier analysis.

OTHER OUTCOMES:
Change in BOLD response to oxygen breathing based on T2 contrast induced by deoxyhemoglobin serving as an endogenous contrast agent | Baseline to day 1 post-SBRT
Change in Kel (washout phase constant) values calculated from the DCE curve | Baseline to day 1 post-SBRT
Change in mean apparent diffusion coefficient generated from diffusion weighted images by using the b values | Baseline to day 1 post-SBRT
Change in miRNA expression | Baseline to up to 3 months
Change in plateau signal intensity calculated from the DCE curve | Baseline to day 1 post-SBRT

CONTACTS AND LOCATIONS:
Overall Officials: Terence Williams, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Sebastian NT, Miller ED, Yang X, Diaz DA, Tan Y, Dowell J, Spain J, Rikabi A, Elliott E, Knopp M, Williams TM. A Pilot Trial Evaluating Stereotactic Body Radiation Therapy to Induce Hyperemia in Combination With Transarterial Chemoembolization for Hepatocellular Carcinoma. Int J Radiat Oncol Biol Phys. 2020 Dec 1;108(5):1276-1283. doi: 10.1016/j.ijrobp.2020.07.033. Epub 2020 Jul 23. PMID 32712254
- See also: The Jamesline — http://cancer.osu.edu